CLINICAL TRIAL: NCT04418466
Title: Open-Label Study in Stable Schizophrenia Patients to Evaluate the Safety, Tolerability, and Pharmacokinetics of Switching From Oral Risperidone to Risperidone Implant (DLP-114)
Brief Title: Safety, Tolerability, and Pharmacokinetics of Switching From Oral Risperidone to Risperidone Implant
Acronym: DLP-114
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Delpor, Inc. (Industry)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DLP-114-03; R44MH094036 (NIH)
Record Dates: First submitted 2020-06-01; First posted 2020-06-05 (Actual); Results first posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Schizophrenia
Keywords: risperidone; schizophrenia; implant
MeSH Terms: conditions — Schizophrenia | interventions — Risperidone

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- DLP-114 alpha-4 (6-months) (Experimental): Group 1: 6-month implant arm Oral phase: 3mg of Risperidone for 2 weeks Implant phase: 2 implants (360mg of Risperidone per implant) for 6 months
  Interventions: Combination Product: Risperidone
- DLP-114 alpha-7 (12-months) (Experimental): Group 2: 12-month implant arm Oral phase: 3mg of Risperidone for 2 weeks Implant phase: 2 implants (435mg of Risperidone per implant) for 12 months
  Interventions: Combination Product: Risperidone

INTERVENTIONS:
Combination Product: Risperidone — Risperidone Implant
  Other Names: DLP-114

SUMMARY:
This is an Open-Label Study in Stable Schizophrenia Patients to Evaluate the Safety, Tolerability, and Pharmacokinetics of Switching from Oral Risperidone to Risperidone Implant (DLP-114).

DETAILED DESCRIPTION:
Phase 1 open-label study in stable schizophrenia patients designed to evaluate the safety, tolerability, and Pharmacokinetics of switching from 2 mg/day or 3 mg/day oral risperidone to two DLP-114 devices for a six or twelve-month dosing period.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients 18-70 years of age of both sexes diagnosed with schizophrenia or schizoaffective disorder according to Diagnostic and Statistical Manual (DSM)-V who have been stable on oral risperidone (2mg-3mg) for at least 2 weeks.
2. Patient (and/or a patient's authorized legal representative) has provided written informed consent
3. Patient meets the following criteria:

   1. Outpatient status
   2. PANSS Total Score ≤ 80 at screening.
   3. A score of ≤ 4 on the following PANSS items:

   i. Conceptual disorganization ii. Suspiciousness iii. Hallucinatory behavior iv. Unusual thought content v. Hostility d. Clinical Global Impression Scale (CGI-S) ≤ 4 (moderately ill)\Lack of clinically significant suicidal ideation or behavior; Columbia Suicide Severity Rating Scale (C-SSRS) score type of 4-5 require evaluation by mental health professional to ensure patient safety in study
4. Body Mass Index (BMI) within the range of 18.5 to 40.0 kg/m2 (inclusive);
5. Ability to understand the nature and objectives of the trial, including risks and adverse events, and be able to read, review and sign the informed consent document prior to conduct of any study procedures;
6. Willing and able to comply with the requirements of the study protocol; including willingness to visit the clinical facility for all outpatient visits and confinement periods;
7. Have suitable venous access for blood sampling.
8. Patient is assessed by the Investigator to be symptomatically stable with regard to pre-existing medical conditions as evidenced by medical history, non-clinically significant findings on physical examination, vital signs, clinical laboratory evaluations (hematology, serum chemistries, and urinalysis) or 12-lead electrocardiogram (ECG). Subjects may continue on their current prescribed medication regimens to control pre-existing medical and psychiatric conditions (other than schizophrenia) including the use of prescribed PRN medications.

Exclusion Criteria:

1. PANSS score at baseline is ≥ 20% change from screening.
2. Hospitalized or required acute crisis intervention for symptom exacerbation in the 60 days prior to admission as determined by the Investigator
3. Patient has a history of suicide attempt in the last year, or in the opinion of the investigator is currently at imminent risk of suicide.
4. Patient experiencing acute depressive symptoms within the past 30 days, according to the Investigator's opinion, that required treatment with an antidepressant
5. Has a current or recent (within 12 months) DSM-V diagnosis of moderate or severe substance use disorder (except for tobacco use disorder) or has a positive urine drug screen for prohibited substances at screening.
6. Have impaired hepatic (Alanine transaminase (ALT) /aspartate aminotransferase (AST) >1.5 times higher than the upper limit of normal) or renal function (eGFR<50 mL/min)
7. Previously defined hypersensitivity to Risperidone
8. History of neuroleptic malignant syndrome (NMS)
9. Electroconvulsive therapy within 6 months of admission
10. Requires current use of agents that are strong inhibitors and inducers of cytochrome P450;
11. Known hypersensitivity or allergy to lidocaine or any local anesthetic agent of the amide type (local anesthetic used during implant and explant procedures);
12. Presence of clinically significant skin disorders (such as, but not limited to, skin cancer, psoriasis, eczema, or atopic dermatitis), evidence of recent sunburn, scar tissue, tattoo, open sore, body piercing or branding at the intended implantation site that would interfere with the implantation procedure or interfere with implant site assessments as determined by the investigator;
13. History of clinically significant hypersensitivity or allergic reactions;
14. Known allergy or hypersensitivity to para-aminobenzoic acid (PABA);
15. Known allergy or hypersensitivity to parabens, local anesthetics of the ester type, and sulfa drugs including antibiotics and thiazide diuretics;
16. Known hypersensitivity to titanium, implant materials or procedure;
17. Administration of an investigational drug or device within 1 month prior to first dosing;
18. Positive result for hepatitis B surface antigen (HBsAg), hepatitis C (HCV) antibody, or HIV antibody;
19. Pregnant or lactating patients. Positive pregnancy test;
20. Positive drug test for Methamphetamines, Opiates, Cocaine, Phencyclidine, Benzodiazepines, Barbiturates, Methadone, Antidepressants and Amphetamines or positive alcohol test at screening or prior to first dose;
21. Poor CYP2D6 metabolizer;
22. History of skin picking or delusional parasitosis;
23. Known history of abnormal scar formation or family history of keloid formation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-02-10 (Actual); Study Completion 2023-02-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Collaborative Neuroscience Research, Long Beach, California
  - Segal Trials, Miami Lakes, Florida

RESULTS

PARTICIPANT FLOW:
Groups:
- DLP-114 Alpha-4 (6-months): Group 1: 6-month implant arm
  Oral Phase: 3mg of Risperidone for 2 weeks
  Implant Phase: 2 implants (360 mg of Risperidone per implant) for 6 months
- DLP-114 Alpha-7 (12-months): Group 2: 12-month implant arm
  Oral Phase: 3 mg of Risperidone for 2 weeks
  Implant Phase: 2 implants (435 mg of Risperidone per implant) for 12 months
Period: Overall Study
Arm/Group | DLP-114 Alpha-4 (6-months) | DLP-114 Alpha-7 (12-months)
Started (Started Oral Phase) | 17 (14 completed the oral phase and started the implant phase.) | 17 (14 completed the oral phase and started the implant phase.)
Started Implant Phase | 14 | 14
Completed (Completed Implant Phase) | 12 (Represents the number that completed the oral and implant phase.) | 11 (Represents the number that completed the oral and implant phase.)
Not Completed | 5 | 6

BASELINE CHARACTERISTICS:
Population: Represents the number of participants who completed the oral phase and enrolled in the implant phase.
Groups:
- DLP-114 Alpha-4 (6-months): Group 1: 6-month implant arm
  Oral Phase: 3 mg of Risperidone for 2 weeks
  Implant Phase: 2 implants (360 mg of Risperidone per implant) for 6 months
- Total: Total of all reporting groups
Arm/Group | DLP-114 Alpha-4 (6-months) | DLP-114 Alpha-7 (12-months) | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 14 | 28
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: Years] | 54.5 [23 to 62] | 54.5 [28 to 64] | 54.5 [23 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 11 | 10 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 12 | 13 | 25
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 13 | 22
  White | 5 | 1 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events
Description: Number of Participants with Treatment-Emergent Adverse Events.
Time Frame: Up to 8 months and up to 15 months for groups 1 and 2 respectively.
Population: All patients participating in both phases of the study (Oral and implant).
Measure: Count of Participants; unit: Participants
Arm/Group | DLP-114 Alpha-4 (6-months) | DLP-114 Alpha-7 (12-months)
Number analyzed (Participants) | 14 | 14
Participants | 10 | 13

2. Primary Outcome: Percentage of Implant Site Assessments With a Dermal Irritation Scale Rating Greater Than Zero
Description: Evaluate the incidence of local site reactions. Percentage of implant site assessments with a dermal irritation scale rating greater than zero (rating scale is 0 to 4, where 0 indicates no erythema or edema, and 4 indicates erythema or slight eschar).
Time Frame: 6 months and 12 months for groups 1 and 2 respectively.
Population: Participants who enrolled in the implant phase of the study,
Measure: Number; unit: percentage of site assessments rated >0
Units Other Than Participants: Implant site assessments
Arm/Group | DLP-114 Alpha-4 (6-months) | DLP-114 Alpha-7 (12-months)
Number analyzed (Participants) | 14 | 14
Number analyzed (Implant site assessments) | 298 | 409
percentage of site assessments rated >0 | 10.1 | 5.1

3. Primary Outcome: Number of Participants Who Experienced an AE Related to Implantation or Explantation Procedures
Description: Number of participants who experienced an Adverse Events related to Implantation or Explantation Procedures
Time Frame: 6 months and 12 months for groups 1 and 2 respectively.
Population: Patients who started the implant phase
Measure: Count of Participants; unit: Participants
Arm/Group | DLP-114 Alpha-4 (6-months) | DLP-114 Alpha-7 (12-months)
Number analyzed (Participants) | 14 | 14
Participants | 7 | 2

4. Secondary Outcome: Oral Phase Cave: Average Plasma Concentration of Active Moiety (Risperidone + 9 OH Risperidone) During 24 Hours After 3 Days of Repeated 3mg QD Oral Administrations
Description: Oral Phase Cave: Average plasma concentration of active moiety (risperidone + 9 OH risperidone) during 24 hours after 3 days of repeated 3mg QD oral administrations
Time Frame: t=0, 0.5, 1, 2, 3, 4, 6, 8, 12, and 24 hours following oral administration.
Population: Participants who completed the Oral Dose Phase and began the Implant Phase.
Measure: Mean (Standard Deviation); unit: ng/mL
Units Other Than Participants: Plasma Measurement
Arm/Group | DLP-114 Alpha-4 (6-months) | DLP-114 Alpha-7 (12-months)
Number analyzed (Participants) | 14 | 14
Number analyzed (Plasma Measurement) | 140 | 140
ng/mL | 43.07 (13.32) | 43.86 (14.12)

5. Secondary Outcome: Implant Cave: Average Plasma Concentration of Active Moiety (Risperidone + 9 OH Risperidone) During the Implant Phase
Description: Average plasma concentration of active moiety (risperidone + 9 OH risperidone) following switch from oral risperidone to subcutaneous implantation of two DLP-114 devices at specific time intervals per protocol for 6 months or 12 months (groups 1 and 2 respectively).
Time Frame: PK blood draw & analysis were performed per protocol time intervals; 0, 1, 2, 3, 4, 6, 8, 12, 24, 28, 32, 36, 48, and 52 hours post-placement of implants; 1x/day for 4 additional days, 1x/week during days 5-28; biweekly until day of device removal.
Population: Participants who completed the study.
Measure: Mean (Standard Deviation); unit: ng/ML
Units Other Than Participants: Plasma Measurement
Arm/Group | DLP-114 Alpha-4 (6-months) | DLP-114 Alpha-7 (12-months)
Number analyzed (Participants) | 12 | 11
Number analyzed (Plasma Measurement) | 361 | 459
ng/ML | 11.54 (3.99) | 14.41 (6.76)

6. Secondary Outcome: Average Positive and Negative Syndrome Scale (PANSS) During the Study (Oral & Implant Phases)
Description: Average Positive and Negative Syndrome Scale (PANSS) during the study (Oral & Implant Phases). The average PANSS score was calculated for each participant during the study. The PANSS score reported is the average of all participants who completed the study in each group. The PANSS provides a total score (sum of the scores of all 30 items) ranging from 30 to 210, higher scores indicate more severe neuropsychiatric symptoms of schizophrenia. Scores for 3 subscales, that is, for positive subscale (sum of the scores of all 7 items) and negative subscale (sum of the scores of all 7 items) ranges from 7 (absent) to 49 (extreme psychopathology), and for the general psychopathology subscale (sum of the scores of all 16 items) score ranges from 16 (absent) to 112 (extreme psychopathology)
Time Frame: For group 1: Screening period, day -1, day 84, day 183; and for Group 2: Screening period, day -1, day 84, day 182, day 280, day 364.
Population: Participants who completed the study.
Measure: Mean (Standard Deviation); unit: Total score on PANSS scale
Units Other Than Participants: Individual PANSS Score Assessment
Arm/Group | DLP-114 Alpha-4 (6-months) | DLP-114 Alpha-7 (12-months)
Number analyzed (Participants) | 12 | 11
Number analyzed (Individual PANSS Score Assessment) | 48 | 66
Total score on PANSS scale | 56.92 (7.55) | 57.51 (8.43)

7. Secondary Outcome: Average Clinical Global Impression-Improvement (CGI-I) Scale During the Implant Phase
Description: Average Clinical Global Impression-Improvement (CGI-I) Scale during the Implant Phase. The average CGI-I score was calculated for each participant during the Implant Phase. The CGI-I score reported is the average of all participants who completed the study in each group. The CGI-I is a 7-point scale that requires the clinician to assess how much the participant's illness has improved or worsened relative to a baseline state at the beginning of the intervention and rated as: 1=very much improved; 2=much improved; 3=minimally improved; 4=no change; 5=minimally worse; 6=much worse; 7=very much worse.
Time Frame: CGI-I assessments were conducted over the course of the study per the protocol schedule of assessments. For Group 1: day 7, 14, 28, 42, 70, 112,140, 68, 183 and for Group 2: day 7, 14, 28, 56, 84, 112,140, 168,182, 210, 238, 252, 280, 308, 336, 350, 364.
Population: Participants who completed the study
Measure: Mean (Full Range); unit: Score on CGI-I scale
Units Other Than Participants: Individual CGI-I Assessment
Arm/Group | DLP-114 Alpha-4 (6-months) | DLP-114 Alpha-7 (12-months)
Number analyzed (Participants) | 12 | 11
Number analyzed (Individual CGI-I Assessment) | 108 | 181
Score on CGI-I scale | 3.5 [1 to 5] | 3.7 [1 to 5]

8. Secondary Outcome: Average Daily Risperidone Implant Output During the Implant Phase
Description: Average daily Risperidone Implant output during the Implant Phase. Average daily output is calculated by using the amount of Risperidone drug substance remaining in the DLP-114 reservoir following removal. The average daily output is calculated for each participant by using the two devices that each participant received. Risperidone output reported as the average for each group.
Time Frame: 6-months and 12-months for groups 1 and 2 respectively. Remaining Risperidone measurements taken at the end of the Implant Phase.
Population: Participants who completed the study.
Measure: Mean (Standard Deviation); unit: mg/day
Units Other Than Participants: Implant Devices
Arm/Group | DLP-114 Alpha-4 (6-months) | DLP-114 Alpha-7 (12-months)
Number analyzed (Participants) | 12 | 11
Number analyzed (Implant Devices) | 24 | 22
mg/day | 0.676 (0.156) | 0.531 (0.106)

9. Secondary Outcome: Implant Device Placement Depth
Description: Average depth of implant device placement measured by ultrasound in mm. The average depth was calculated for each participant. The implant device depth reported is the average of all participants who completed the study in each group.
Time Frame: Group 1 (6-month): Ultrasound on days 14 and 183. Group 2 (12-month): Ultrasound on days 14 and 364.
Population: Participants who completed the study
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Implant Devices
Arm/Group | DLP-114 Alpha-4 (6-months) | DLP-114 Alpha-7 (12-months)
Number analyzed (Participants) | 12 | 11
Number analyzed (Implant Devices) | 24 | 22
mm | 4.10 (1.84) | 4.85 (1.40)

10. Secondary Outcome: Number of Participants Who Experienced Implant Migration in at Least One of the Implanted Devices
Description: Implant migration is defined as a distance of greater than 3cm between the initial incision and the proximal end of the implant device prior to removal.
Time Frame: Group 1 (6-month): Assessments performed day 1 and day 183. Group 2 (12-month): Assessments performed day 1 and 364.
Population: Participants who completed the study.
Measure: Number; unit: number of participants
Arm/Group | DLP-114 Alpha-4 (6-months) | DLP-114 Alpha-7 (12-months)
Number analyzed (Participants) | 12 | 11
number of participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Group 1 (6-month implant group): Up to 8-months (Includes oral phase, implant phase, and follow up). Group 2 (12-month implant group): Up to 15-months (Includes oral phase, implant phase, and follow up).
Groups:
- DLP-114 Alpha-4 (6-months): 2 360mg Risperidone Implants
  Risperidone: Risperidone Implant
- DLP-114 Alpha-7 (12-months): 2 435mg Risperidone Implants
  Risperidone: Risperidone Implant
Arm/Group | DLP-114 Alpha-4 (6-months) | DLP-114 Alpha-7 (12-months)
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 1/14
Other Adverse Events (participants affected / at risk) | 10/14 | 12/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DLP-114 Alpha-4 (6-months) (N=14) | DLP-114 Alpha-7 (12-months) (N=14)
Oedema Peripheral (General disorders) | 0 (0) | 1 (1)
Weight Increase (Investigations) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cardiac Failure Congestive (Cardiac disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DLP-114 Alpha-4 (6-months) (N=14) | DLP-114 Alpha-7 (12-months) (N=14)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Implant site haemorrhage (General disorders) | 1 (2) | 0 (0)
Injection Site Scar (General disorders) | 1 (2) | 0 (0)
Implant site pain (General disorders) | 2 (3) | 2 (4)
Insomnia (Psychiatric disorders) | 1 (2) | 3 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0)
Somnolence (Nervous system disorders) | 2 (3) | 1 (1)
Chest Pain (General disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (3) | 1 (2)
Vomiting (Gastrointestinal disorders) | 1 (3) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Weight increased (Investigations) | 3 (5) | 0 (0)
Implant Site pruritus (General disorders) | 1 (1) | 0 (0)
Ankle Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Injection site discomfort (General disorders) | 0 (0) | 2 (4)
Paresthesia Oral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal Discomfort (Gastrointestinal disorders) | 1 (3) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (3) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (2) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Ear infection (Infections and infestations) | 1 (2) | 0 (0)
Abnormal behavior (Psychiatric disorders) | 1 (3) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (3) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (3) | 0 (0)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (3) | 0 (0)
Polycythaemia (Blood and lymphatic system disorders) | 1 (3) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (3) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (3) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (2) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Ligament Sprain (Injury, poisoning and procedural complications) | 1 (3) | 0 (0)
Testicular pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3)
Hordeolum (Infections and infestations) | 1 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (3):
  • Study Protocol (2021-07-12): https://cdn.clinicaltrials.gov/large-docs/66/NCT04418466/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-20): https://cdn.clinicaltrials.gov/large-docs/66/NCT04418466/SAP_001.pdf
  • Informed Consent Form (2021-09-21): https://cdn.clinicaltrials.gov/large-docs/66/NCT04418466/ICF_002.pdf